CLINICAL TRIAL: NCT00223080
Title: A Phase III Trial of Aventis Pasteur Live Recombinant ALVAC-HIV (vCP1521) Priming With VaxGen gp120 B/E (AIDSVAX B/E) Boosting in HIV-uninfected Thai Adults
Brief Title: HIV Vaccine Trial in Thai Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: United States Army Medical Materiel Development Activity (U.S. Federal Agency); Armed Forces Research Institute of Medical Sciences, Thailand (Other Government); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); MCM Vaccines B.V. (Industry); VaxGen (Industry); The Emmes Company, LLC (Industry); Ministry of Health, Thailand (Other Government); Mahidol University (Other); Royal Thai Army Medical Department (Other Government); Tripler Army Medical Center (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RV144; HSRRB A-11048 (Other: USAMRMC HSRRB)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: HIV Infection
Keywords: HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine (Active Comparator): ALVAC-HIV vCP1521 + AIDSVAX will both be administered by the intramuscular route (preferably in the deltoid region) on weeks 0, 4, 12, and 24.
  Interventions: Biological: ALVAC-HIV vCP1521 + AIDSVAX
- Placebo (Placebo Comparator): ALVAC Placebo + AIDSVAX Placebo will be administered at week 12 and 24. ALVAC Placebo only was additionally administered at week 0 and 4.
  Interventions: Other: ALVAC Placebo + AIDSVAX Placebo

INTERVENTIONS:
Biological: ALVAC-HIV vCP1521 + AIDSVAX — Combined dose of 600 μg (300 μg of each antigen), co-formulated and administered in alumi-um hydroxide gel at a dose of 600 μg/mL
  Other Names: ALVAC-HIV (vCP1521) >106 CCID50 per 1 mL dose; AIDSVAX® B/E; Bivalent HIV gp120 vaccine subtype B (MN), and E (A244)
  Arms: Vaccine
Other: ALVAC Placebo + AIDSVAX Placebo — ALVAC carrier, supplied as a lyophilized product, without virus and Aluminum hydroxide adjuvant, 1.2 mL per vial, given as a 1 mL injection
  Other Names: ALVAC carrier lyophilized product without virus; Aluminum hydroxide adjuvant
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether immunizations with an integrated combination of ALVAC-HIV (vCP1521) boosted by AIDSVAX gp120 B/E prevent HIV infection in healthy Thai volunteers.

DETAILED DESCRIPTION:
A vaccine for the prevention of HIV infection remains an urgent need as part of the efforts to control the HIV pandemic. In this phase III efficacy trial, a 'prime-boost' vaccine strategy is evaluated for prevention of infection and amelioration of disease course. ALVAC-HIV (vCP1521) from sanofi pasteur is given as the 'prime' vaccine at months 0, 1, 3 and 6; AIDSVAX gp120 B/E from VaxGen is given as the 'boost' at months 3 and 6. This regimen will be given to 8,000 adult Thai subjects, while another 8,000 will be given placebos in a double-blinded, randomized manner. Following the completion of each subjects immunization phase, he/she will be followed for 3 years with clinic visits every 6 months with HIV testing, pre- and post-test counseling. Subjects who become HIV infected will be counseled, referred to HIV treatment facilities for management according to national guidelines, and offered enrollment in a protocol for extended follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Possession of the 13-digit Thai National ID card
* 18-30 years of age (inclusive), male or female
* For women, a negative urine pregnancy test on the day of enrollment, as well as assurance that adequate birth control measures would be applied during the course of the injections and the 3 months after the last injection.
* Absence of systemic disease or immunodeficiency as determined by medical history and directed physical examination.
* Negative serology for HIV-1 infection within 45 days prior to enrollment.
* Availability and commitment for 3.5 years of participation.
* Able to understand the study (shown by receiving a passing score on the Test of Understanding administered under the screening protocol) and gave written informed consent.
* Enrollment in and referral from screening protocol, RV148

Exclusion Criteria:

* Previous participation in any HIV vaccine trial (unless the volunteer could provide documentation that he/she received placebo).
* Active tuberculosis, other systemic disease process, or immunodeficiency as detected by medical history and directed physical examination that would, in the opinion of the investigator, impede compliance with study requirements or complicate the interpretation of adverse events.
* Any significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study or might interfere with the volunteer's ability to successfully complete the study.
* Occupational or other responsibilities that would prevent completion of 3.5 years of participation in the study.
* History of anaphylaxis or other serious adverse reactions to vaccines, or allergies or reactions likely to be exacerbated by any component of the vaccine or placebo, including egg products and neomycin.
* Women breast-feeding or pregnant (positive pregnancy test) or planning to become pregnant during the 9-month window between study enrollment and 3-months after the last vaccination visit.
* Study site employees who were involved in the protocol and may have had direct access to trial-related data.
* Chronic use of therapies which may modify immune response, such as IV immune globulin and systemic corticosteroids (in doses of > 20 mg prednisone equivalent for periods exceeding 10 days), and use of experimental drugs or vaccines.
* Receipt of a non-HIV vaccine or immune globulins within 14 days.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16402 (Actual)
Dates: Start 2003-10; Primary Completion 2006-07 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Supachai Rerks-Ngarm, MD, Principal Investigator — Ministry of Health, Thailand
Locations (8):
- Thailand (8):
  - Ban Lamung District Hospital, Ban Lamung District, Changwat Chon Buri
  - Phan Tong District Hospital, Phan Tong District, Changwat Chon Buri
  - Sattahip District Hospital, Sattahip District, Changwat Chon Buri
  - Ao Udom Hospital, Sri Racha District, Changwat Chon Buri
  - Ban Chang District Hospital, Ban Chang District, Changwat Rayong
  - Ban Khai District Hospital, Ban Khai District, Changwat Rayong
  - Klaeng District Hospital, Klaeng District, Changwat Rayong
  - Provincial Health Office, Muang District, Changwat Rayong

REFERENCES:
- [Background] Nitayaphan S, Pitisuttithum P, Karnasuta C, Eamsila C, de Souza M, Morgan P, Polonis V, Benenson M, VanCott T, Ratto-Kim S, Kim J, Thapinta D, Garner R, Bussaratid V, Singharaj P, el-Habib R, Gurunathan S, Heyward W, Birx D, McNeil J, Brown AE; Thai AIDS Vaccine Evaluation Group. Safety and immunogenicity of an HIV subtype B and E prime-boost vaccine combination in HIV-negative Thai adults. J Infect Dis. 2004 Aug 15;190(4):702-6. doi: 10.1086/422258. Epub 2004 Jul 20. PMID 15272397
- [Background] Karnasuta C, Paris RM, Cox JH, Nitayaphan S, Pitisuttithum P, Thongcharoen P, Brown AE, Gurunathan S, Tartaglia J, Heyward WL, McNeil JG, Birx DL, de Souza MS; Thai AIDS Vaccine Evaluation Group, Thailand. Antibody-dependent cell-mediated cytotoxic responses in participants enrolled in a phase I/II ALVAC-HIV/AIDSVAX B/E prime-boost HIV-1 vaccine trial in Thailand. Vaccine. 2005 Mar 31;23(19):2522-9. doi: 10.1016/j.vaccine.2004.10.028. PMID 15752839
- [Background] Brown AE, Nitayaphan S. Foundations for a Phase III human immunodeficiency virus vaccine trial: A decade of Thai-U.S. Army collaborative research. Mil Med. 2004 Aug;169(8):588-93. doi: 10.7205/milmed.169.8.588. PMID 15379068
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Williams LD, Shen X, Sawant SS, Akapirat S, Dahora LC, Tay MZ, Stanfield-Oakley S, Wills S, Goodman D, Tenney D, Spreng RL, Zhang L, Yates NL, Montefiori DC, Eller MA, Easterhoff D, Hope TJ, Rerks-Ngarm S, Pittisuttithum P, Nitayaphan S, Excler JL, Kim JH, Michael NL, Robb ML, O'Connell RJ, Karasavvas N, Vasan S, Ferrari G, Tomaras GD; RV305 study team. Viral vector delivered immunogen focuses HIV-1 antibody specificity and increases durability of the circulating antibody recall response. PLoS Pathog. 2023 May 31;19(5):e1011359. doi: 10.1371/journal.ppat.1011359. eCollection 2023 May. PMID 37256916
- [Derived] Zhao LP, Fiore-Gartland A, Carpp LN, Cohen KW, Rouphael N, Fleurs L, Dintwe O, Zhao M, Moodie Z, Fong Y, Garrett N, Huang Y, Innes C, Janes HE, Lazarus E, Michael NL, Nitayaphan S, Pitisuttithum P, Rerks-Ngarm S, Robb ML, De Rosa SC, Corey L, Gray GE, Seaton KE, Yates NL, McElrath MJ, Frahm N, Tomaras GD, Gilbert PB. Landscapes of binding antibody and T-cell responses to pox-protein HIV vaccines in Thais and South Africans. PLoS One. 2020 Jan 30;15(1):e0226803. doi: 10.1371/journal.pone.0226803. eCollection 2020. PMID 31999736
- [Derived] Akapirat S, Karnasuta C, Vasan S, Rerks-Ngarm S, Pitisuttithum P, Madnote S, Savadsuk H, Rittiroongrad S, Puangkaew J, Phogat S, Tartaglia J, Sinangil F, de Souza MS, Excler JL, Kim JH, Robb ML, Michael NL, Ngauy V, O'Connell RJ, Karasavvas N; RV305 Study Group. Characterization of HIV-1 gp120 antibody specificities induced in anogenital secretions of RV144 vaccine recipients after late boost immunizations. PLoS One. 2018 Apr 27;13(4):e0196397. doi: 10.1371/journal.pone.0196397. eCollection 2018. PMID 29702672
- [Derived] Huang Y, Zhang L, Janes H, Frahm N, Isaacs A, Kim JH, Montefiori D, McElrath MJ, Tomaras GD, Gilbert PB. Predictors of durable immune responses six months after the last vaccination in preventive HIV vaccine trials. Vaccine. 2017 Feb 22;35(8):1184-1193. doi: 10.1016/j.vaccine.2016.09.053. Epub 2017 Jan 25. PMID 28131393
- [Derived] Dommaraju K, Kijak G, Carlson JM, Larsen BB, Tovanabutra S, Geraghty DE, Deng W, Maust BS, Edlefsen PT, Sanders-Buell E, Ratto-Kim S, deSouza MS, Rerks-Ngarm S, Nitayaphan S, Pitisuttihum P, Kaewkungwal J, O'Connell RJ, Robb ML, Michael NL, Mullins JI, Kim JH, Rolland M. CD8 and CD4 epitope predictions in RV144: no strong evidence of a T-cell driven sieve effect in HIV-1 breakthrough sequences from trial participants. PLoS One. 2014 Oct 28;9(10):e111334. doi: 10.1371/journal.pone.0111334. eCollection 2014. PMID 25350851
- [Derived] Gartland AJ, Li S, McNevin J, Tomaras GD, Gottardo R, Janes H, Fong Y, Morris D, Geraghty DE, Kijak GH, Edlefsen PT, Frahm N, Larsen BB, Tovanabutra S, Sanders-Buell E, deCamp AC, Magaret CA, Ahmed H, Goodridge JP, Chen L, Konopa P, Nariya S, Stoddard JN, Wong K, Zhao H, Deng W, Maust BS, Bose M, Howell S, Bates A, Lazzaro M, O'Sullivan A, Lei E, Bradfield A, Ibitamuno G, Assawadarachai V, O'Connell RJ, deSouza MS, Nitayaphan S, Rerks-Ngarm S, Robb ML, Sidney J, Sette A, Zolla-Pazner S, Montefiori D, McElrath MJ, Mullins JI, Kim JH, Gilbert PB, Hertz T. Analysis of HLA A*02 association with vaccine efficacy in the RV144 HIV-1 vaccine trial. J Virol. 2014 Aug;88(15):8242-55. doi: 10.1128/JVI.01164-14. Epub 2014 May 14. PMID 24829343
- [Derived] Zolla-Pazner S, deCamp A, Gilbert PB, Williams C, Yates NL, Williams WT, Howington R, Fong Y, Morris DE, Soderberg KA, Irene C, Reichman C, Pinter A, Parks R, Pitisuttithum P, Kaewkungwal J, Rerks-Ngarm S, Nitayaphan S, Andrews C, O'Connell RJ, Yang ZY, Nabel GJ, Kim JH, Michael NL, Montefiori DC, Liao HX, Haynes BF, Tomaras GD. Vaccine-induced IgG antibodies to V1V2 regions of multiple HIV-1 subtypes correlate with decreased risk of HIV-1 infection. PLoS One. 2014 Feb 4;9(2):e87572. doi: 10.1371/journal.pone.0087572. eCollection 2014. PMID 24504509
- [Derived] Pitisuttithum P, Rerks-Ngarm S, Bussaratid V, Dhitavat J, Maekanantawat W, Pungpak S, Suntharasamai P, Vanijanonta S, Nitayapan S, Kaewkungwal J, Benenson M, Morgan P, O'Connell RJ, Berenberg J, Gurunathan S, Francis DP, Paris R, Chiu J, Stablein D, Michael NL, Excler JL, Robb ML, Kim JH. Safety and reactogenicity of canarypox ALVAC-HIV (vCP1521) and HIV-1 gp120 AIDSVAX B/E vaccination in an efficacy trial in Thailand. PLoS One. 2011;6(12):e27837. doi: 10.1371/journal.pone.0027837. Epub 2011 Dec 21. PMID 22205930
- [Derived] Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Kaewkungwal J, Chiu J, Paris R, Premsri N, Namwat C, de Souza M, Adams E, Benenson M, Gurunathan S, Tartaglia J, McNeil JG, Francis DP, Stablein D, Birx DL, Chunsuttiwat S, Khamboonruang C, Thongcharoen P, Robb ML, Michael NL, Kunasol P, Kim JH; MOPH-TAVEG Investigators. Vaccination with ALVAC and AIDSVAX to prevent HIV-1 infection in Thailand. N Engl J Med. 2009 Dec 3;361(23):2209-20. doi: 10.1056/NEJMoa0908492. Epub 2009 Oct 20. PMID 19843557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16,402 subjects were randomized, 16,395 were infection free and assigned treatment groups
Pre-assignment Details: 16,402 individuals were randomly assigned to the 2 treatment arms. 7 individuals were identified as having human immunodeficiency virus (HIV) infection that was present pre-vaccination detected by polymerase chain reaction (PCR) amplification. These individuals were removed from the modified intent to treat (MITT) population.
Period: Overall Study
Arm/Group | Vaccine | Placebo
Started | 8197 | 8198
Completed | 7401 | 7401
Not Completed | 796 | 797
Not completed — Withdrawal by Subject | 253 | 232
Not completed — Required contraindicated med | 0 | 1
Not completed — Non-compliant | 7 | 7
Not completed — Moved from study area | 37 | 47
Not completed — Lost to Follow-up | 259 | 284
Not completed — Death | 85 | 74
Not completed — Other | 14 | 11
Not completed — Reason not provided | 141 | 140
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (MITT) Population - those participants who were infection free at entry into the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Total
Number analyzed (Participants) | 8197 | 8198 | 16395
Age, Customized [Count of Participants; unit: Participants]
  18 - 20 | 2297 | 2246 | 4543
  21 - 25 | 3633 | 3708 | 7341
  26 - 30 | 2267 | 2244 | 4511
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3164 | 3167 | 6331
  Male | 5033 | 5031 | 10064
Province [Number; unit: participants]
  Chon Buri | 4107 | 4107 | 8214
  Rayong | 4090 | 4091 | 8181
Marital status [Number; unit: participants]
  Single | 3353 | 3338 | 6691
  Married | 4110 | 4169 | 8279
  Divorced | 602 | 541 | 1143
  Widowed | 50 | 64 | 114
  Separated | 82 | 86 | 168
Number of sex partners [Number; unit: participants]
  0 | 1864 | 1801 | 3665
  1 | 5428 | 5495 | 10923
  > 1 | 619 | 620 | 1239
  Did not answer | 280 | 273 | 553
  Missing data | 6 | 9 | 15
Risk group [Number; unit: participants]
  Low | 3865 | 3924 | 7789
  Medium | 2369 | 2292 | 4661
  High | 1963 | 1982 | 3945

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of HIV-1 Infection Rate in Intent to Treat Population
Description: HIV-1 infection rate. Detection of HIV-1 infection was defined according to the HIV diagnostic algorithm utilizing serologic and nucleic acid technologies. Incidence of HIV infection was compared in the vaccine and placebo-recipient groups.
Time Frame: 42 Months
Population: Modified Intent-to-Treat (MITT) Population: those participants who were infection free at entry into the study
Measure: Number (95% Confidence Interval); unit: Percetage of subjects
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 8197 | 8198
Percetage of subjects
  12 months | 0.15 [0.07 to 0.24] | 0.38 [0.24 to 0.52]
  24 months | 0.41 [0.27 to 0.55] | 0.64 [0.46 to 0.82]
  36 months | 0.58 [0.41 to 0.75] | 0.84 [0.63 to 1.04]
  42 months | 0.68 [0.49 to 0.87] | 0.96 [0.74 to 1.18]

2. Primary Outcome: Vaccine Efficacy as Determined by Acquisition of Infection in the Per-protocol Population
Description: Cumulative Number of HIV Infections. Detection of HIV-1 infection was defined according to the HIV diagnostic algorithm utilizing serologic and nucleic acid technologies. Incidence of HIV infection was compared in the vaccine and placebo-recipient groups.
Time Frame: 42 Months
Population: Per-protocol population: The per-protocol analysis is restricted to the individuals who were infection-free at the completion of vaccination and who received a timely set of 4 vaccinations.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 6176 | 6366
Percentage of subjects
  12 months | 0.08 [0.01 to 0.15] | 0.25 [0.13 to 0.38]
  24 months | 0.36 [0.21 to 0.51] | 0.49 [0.32 to 0.66]
  36 months | 0.52 [0.34 to 0.71] | 0.70 [0.49 to 0.91]
  42 months | 0.59 [0.40 to 0.78] | 0.80 [0.58 to 1.02]

3. Secondary Outcome: Changes in CD4 T Cell Count in Volunteers Who Developed HIV Infection During the Trial for MITT Population
Description: Two CD4 cell counts were obtained (at the verification blood draw and the notification blood draw) and through the remainder of the follow-up period. Results were compared in vaccine and placebo recipients who became HIV-infected during the trial.
Time Frame: 42 weeks
Population: Prior to the analysis, the SAP identified the MITT as those participants who were infection free at entry into the study. Although individuals were screened for HIV antibody prior to entry, individuals identified by laboratory examination of PCR assessments of blinded pre-randomization specimens that were performed subsequent to entry were excluded
Measure: Mean (Standard Error); unit: cells / µL
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 51 | 73
cells / µL
  1st verification | 565.4 (43.5) | 566.7 (26.5)
  Notification | 539.6 (37.1) | 570.6 (29.2)

4. Primary Outcome: Changes in HIV-1 Viral Load in Volunteers Developing HIV Infection During the Trial for the MITT Population
Description: Log10 HIV-1 viral loads for diagnostic specimens for subjects with post-HIV infection. The trial quantitated HIV plasma viral load at the time of diagnosis and through the remainder of the follow-up period. Peri infection results were compared in vaccine and placebo recipients who became HIV-infected during the trial.
Time Frame: 42 months
Population: Modified Intent-to-Treat (MITT) Population: those participants who were infection free at entry into the study
Measure: Mean (Standard Error); unit: log [HIV-1 viral load (unitless)]
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 51 | 73
log [HIV-1 viral load (unitless)]
  First positive serology | 4.379 (0.127) | 4.187 (0.101)
  3-weeks post identificaiton | 4.229 (0.130) | 4.235 (0.095)
  ~6-weeks post identification | 4.274 (0.125) | 4.167 (0.104)

5. Primary Outcome: Changes in HIV-1 Viral Load in Volunteers Developing HIV Infection During the Trial for the Per Protocol Population
Description: as for outcome 4
Time Frame: 42 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log [HIV-1 viral load (unitless)]
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 36 | 50
log [HIV-1 viral load (unitless)]
  First positive serology | 4.307 (0.154) | 4.153 (0.136)
  3-weeks post identificaiton | 4.128 (0.161) | 4.276 (0.118)
  ~6-weeks post identification | 4.280 (0.152) | 4.143 (0.143)

6. Secondary Outcome: Safety Assessment (SAE's and AEs)
Description: The intent-to-treat population is used for analysis of AEs and treatment emergent events are reported. Participant AE rates for all AEs, SAEs and treatment-related AEs are summarized
Time Frame: Dose Interval 1: week 0, Dose Interval 2: Week 4, Dose Interval 3: Week 12, and Dose Interval 4: Week 24; every 6 months during 3 year f/u period
Population: intent-to-treat population
Measure: Number; unit: adverse events
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 8197 | 8198
adverse events
  30-day post dose interval 1 | 1277 | 1336
  30-day post dose interval 2 | 816 | 860
  30-day post dose interval 3 | 614 | 597
  30-day post dose interval 4 | 599 | 630
  All treatment emergent | 5627 | 5685

7. Secondary Outcome: Change in HIV Risk Behaviors Associated With Participation in the Vaccine Trial (MITT)
Description: Self Report of Risk Behavior Status by Treatment and Time. Specifically, this is the responses to the question "Do you think that your everyday behavior puts you at risk for HIV infection?" Modified intent to treat population (MITT)
Time Frame: Week 182
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 7399 | 7395
participants
  Yes | 702 | 763
  No | 6223 | 6130
  Don't know/Not sure | 473 | 502
  Missing value | 1 | 0

ADVERSE EVENTS:
Time Frame: For serious adverse events - anytime after the first vaccination until final follow-up at week 184. For other adverse events - total post-injection reaction severity
Arm/Group | Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 85/8197 | 75/8198
Serious Adverse Events (participants affected / at risk) | 1175/8197 | 1219/8198
Other Adverse Events (participants affected / at risk) | 7442/8197 | 6141/8198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=8197) | Placebo (N=8198)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 1
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 2
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiomegaly (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 1
Extrasystoles (Cardiac disorders) | 2 | 2
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 2 | 0
Cleft lip (Congenital, familial and genetic disorders) | 1 | 0
Cleft lip and palate (Congenital, familial and genetic disorders) | 1 | 0
Cleft palate (Congenital, familial and genetic disorders) | 0 | 1
Congenital anomaly (Congenital, familial and genetic disorders) | 2 | 0
Congenital heart valve disorder (Congenital, familial and genetic disorders) | 1 | 0
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 1 | 0
Congenital megacolon (Congenital, familial and genetic disorders) | 1 | 0
Congenital skin disorder (Congenital, familial and genetic disorders) | 0 | 1
Ebstein's anomaly (Congenital, familial and genetic disorders) | 1 | 0
Familial periodic paralysis (Congenital, familial and genetic disorders) | 0 | 1
Foetal cystic hygroma (Congenital, familial and genetic disorders) | 1 | 0
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 5 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Limb malformation (Congenital, familial and genetic disorders) | 0 | 1
Multiple congenital abnormalities (Congenital, familial and genetic disorders) | 0 | 1
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 | 0
Polydactyly (Congenital, familial and genetic disorders) | 0 | 2
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 | 0
Transposition of the great vessels (Congenital, familial and genetic disorders) | 1 | 0
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 1
Urachal abnormality (Congenital, familial and genetic disorders) | 1 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 2 | 2
Auricular perichondritis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 2
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 0
Thyrotoxic crisis (Endocrine disorders) | 1 | 0
Thyrotoxic periodic paralysis (Endocrine disorders) | 1 | 0
Photokeratitis (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 2 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 7
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal polyp (Gastrointestinal disorders) | 0 | 1
Appendicitis perforated (Gastrointestinal disorders) | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 8 | 12
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 13 | 15
Enteritis (Gastrointestinal disorders) | 4 | 3
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 4 | 2
Gastritis (Gastrointestinal disorders) | 10 | 14
Gastritis alcoholic (Gastrointestinal disorders) | 0 | 1
Gastritis alcoholic haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 3
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 10 | 10
Inguinal hernia, obstructive (Gastrointestinal disorders) | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 6 | 8
Peptic ulcer perforation (Gastrointestinal disorders) | 4 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 6
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Drowning (General disorders) | 1 | 4
Electrocution (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 0
Foreign body reaction (General disorders) | 1 | 0
Lipogranuloma (General disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 14
Sudden death (General disorders) | 0 | 1
Cholangitis acute (General disorders) | 1 | 0
Cholecystitis acute (General disorders) | 2 | 0
Cholecystitis chronic (General disorders) | 1 | 0
Cholelithiasis (General disorders) | 1 | 0
Gallbladder polyp (General disorders) | 1 | 0
Hepatitis (General disorders) | 2 | 2
Hepatitis alcoholic (General disorders) | 0 | 2
Hepatitis fulminant (General disorders) | 0 | 1
Jaundice cholestatic (General disorders) | 0 | 1
Post cholecystectomy syndrome (General disorders) | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 1
Allergy to arthropod sting (Immune system disorders) | 1 | 4
Anaphylactic reaction (Immune system disorders) | 4 | 4
Anaphylactic shock (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 1
Food allergy (Immune system disorders) | 1 | 2
Immune reconstitution syndrome (Immune system disorders) | 1 | 0
Abortion infected (Infections and infestations) | 1 | 2
Abscess (Infections and infestations) | 0 | 1
Abscess jaw (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 2 | 2
Abscess neck (Infections and infestations) | 0 | 1
Abscess oral (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 1
Acute tonsillitis (Infections and infestations) | 6 | 10
Amoebic dysentery (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 3 | 1
Anogenital warts (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 54 | 61
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial labyrinthitis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bartholin's abscess (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 7 | 11
Cellulitis (Infections and infestations) | 4 | 6
Chronic tonsillitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 2 | 3
Dengue fever (Infections and infestations) | 57 | 45
Dermatitis infected (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 4 | 2
Disseminated tuberculosis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Endometritis (Infections and infestations) | 1 | 0
Endometritis decidual (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 19 | 22
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Giardiasis (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 2 | 0
Hepatitis B (Infections and infestations) | 4 | 3
Hepatitis viral (Infections and infestations) | 0 | 1
Hookworm infection (Infections and infestations) | 1 | 0
Infected bites (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 3 | 1
Infection in an immunocompromised host (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 11
Leptospirosis (Infections and infestations) | 1 | 2
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Lymph node tuberculosis (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 4 | 2
Measles (Infections and infestations) | 4 | 2
Meningitis (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0
Meningitis tuberculous (Infections and infestations) | 1 | 1
Meningitis viral (Infections and infestations) | 2 | 0
Mumps (Infections and infestations) | 1 | 0
Murine typhus (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Orchitis (Infections and infestations) | 2 | 2
Osteomyelitis (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 4 | 0
Paronychia (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 14 | 12
Perineal infection (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 24 | 20
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 4 | 2
Plasmodium falciparum infection (Infections and infestations) | 1 | 3
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 10 | 9
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pneumonia measles (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 3
Postoperative wound infection (Infections and infestations) | 3 | 3
Pulmonary tuberculosis (Infections and infestations) | 2 | 4
Pyelonephritis (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 14 | 26
Pyomyositis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Rickettsiosis (Infections and infestations) | 1 | 0
Rubella (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Salpingitis (Infections and infestations) | 0 | 2
Scrub typhus (Infections and infestations) | 4 | 1
Sepsis (Infections and infestations) | 5 | 4
Sialoadenitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 11 | 7
Tooth abscess (Infections and infestations) | 2 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 1 | 1
Typhoid fever (Infections and infestations) | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 15
Urinary tract infection (Infections and infestations) | 14 | 16
Vaginal cellulitis (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 10 | 13
Viral skin infection (Infections and infestations) | 2 | 2
Wound infection (Infections and infestations) | 5 | 8
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 24 | 22
Accident at home (Injury, poisoning and procedural complications) | 1 | 0
Accident at work (Injury, poisoning and procedural complications) | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 2
Animal bite (Injury, poisoning and procedural complications) | 2 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 2
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 3
Cataract traumatic (Injury, poisoning and procedural complications) | 1 | 1
Caustic injury (Injury, poisoning and procedural complications) | 1 | 2
Chemical eye injury (Injury, poisoning and procedural complications) | 1 | 0
Chemical injury (Injury, poisoning and procedural complications) | 0 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 5
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 6 | 6
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Crushing injury of trunk (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Electric shock (Injury, poisoning and procedural complications) | 1 | 1
Exposure to toxic agent (Injury, poisoning and procedural complications) | 2 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Eye penetration (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 3 | 4
Fall (Injury, poisoning and procedural complications) | 14 | 7
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 2
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 20 | 21
Hand fracture (Injury, poisoning and procedural complications) | 2 | 4
Head injury (Injury, poisoning and procedural complications) | 4 | 6
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Induced abortion haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 6 | 15
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 2 | 4
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 3 | 3
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 2
Limb traumatic amputation (Injury, poisoning and procedural complications) | 2 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 9 | 12
Muscle injury (Injury, poisoning and procedural complications) | 2 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 3
Near drowning (Injury, poisoning and procedural complications) | 0 | 1
Open fracture (Injury, poisoning and procedural complications) | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 2 | 2
Overdose (Injury, poisoning and procedural complications) | 6 | 7
Penetrating abdominal trauma (Infections and infestations) | 1 | 0
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Poisoning deliberate (Infections and infestations) | 2 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 5
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 322 | 318
Sciatic nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 3 | 5
Skull fracture (Injury, poisoning and procedural complications) | 1 | 2
Snake bite (Injury, poisoning and procedural complications) | 9 | 8
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Sports injury (Injury, poisoning and procedural complications) | 3 | 4
Tendon injury (Injury, poisoning and procedural complications) | 2 | 3
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Testicular injury (Infections and infestations) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 2 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 | 2
Traumatic shock (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Infections and infestations) | 4 | 2
Urinary bladder rupture (Infections and infestations) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
Gestational diabetes (Metabolism and nutrition disorders) | 0 | 3
Glucose tolerance impaired in pregnancy (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spondylolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angiocentric lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Alcoholic seizure (Nervous system disorders) | 3 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1
Demyelination (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 2
Encephalitis (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 2 | 2
Grand mal convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 3
Migraine (Nervous system disorders) | 5 | 3
Myelitis transverse (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Post-traumatic epilepsy (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 3 | 2
Tension headache (Nervous system disorders) | 4 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vascular headache (Nervous system disorders) | 0 | 2
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 10 | 16
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 13 | 10
Abortion incomplete complicated (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 3 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 73 | 54
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 4 | 4
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 6 | 7
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 12
False labour (Pregnancy, puerperium and perinatal conditions) | 2 | 4
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Foetal growth retardation (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Hydrops foetalis (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 10 | 13
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Labour complication (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 5 | 5
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Post abortion haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 5 | 7
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 12 | 12
Pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 6 | 5
Premature labour (Pregnancy, puerperium and perinatal conditions) | 5 | 3
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 5 | 12
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 3 | 4
Third stage postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 6 | 9
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 2
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 2
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Completed suicide (Psychiatric disorders) | 10 | 6
Depression (Psychiatric disorders) | 0 | 2
Major depression (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1
Schizophrenia (Psychiatric disorders) | 1 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 3
Suicide attempt (Psychiatric disorders) | 24 | 23
Calculus bladder (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 4 | 2
Calculus urinary (Renal and urinary disorders) | 2 | 0
Nephrotic syndrome (Renal and urinary disorders) | 3 | 3
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 2
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Stag horn calculus (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 2
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 2 | 2
Ovarian cyst ruptured (Reproductive system and breast disorders) | 3 | 3
Ovarian cyst torsion (Reproductive system and breast disorders) | 3 | 0
Ovarian mass (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Varicocele (Reproductive system and breast disorders) | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigus (Skin and subcutaneous tissue disorders) | 1 | 0
Pityriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 2
Physical assault (Social circumstances) | 0 | 1
Abortion induced (Surgical and medical procedures) | 3 | 5
Caesarean section (Surgical and medical procedures) | 0 | 1
Endometriosis ablation (Surgical and medical procedures) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3.3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=8197) | Placebo (N=8198)
Headache (General disorders) | 3677 | 2522
Fatigue (General disorders) | 5182 | 3410
Nausea/Vomiting (General disorders) | 1030 | 802
Myalgia (General disorders) | 4237 | 2494
Arthralgia (General disorders) | 2177 | 1246
Rash (Skin and subcutaneous tissue disorders) | 266 | 273
Oral Temperature (General disorders) | 1564 | 1009
Pain/Tenderness (General disorders) | 6852 | 3727 — Local left (ALVAC)
Swelling (General disorders) | 2325 | 432 — Local left (ALVAC)
Arm Movement Limitation (General disorders) | 5647 | 2129 — Local left (ALVAC)
Induration (General disorders) | 316 | 108 — Local left (ALVAC)
Erythema (General disorders) | 283 | 177 — Local left (ALVAC)
Pain/Tenderness (General disorders) | 3543 | 2991 — Local right (AIDSVAX)
Swelling (General disorders) | 643 | 379 — Local right (AIDSVAX)
Arm Movement Limitation (General disorders) | 2627 | 1943 — Local right (AIDSVAX)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No